CLINICAL TRIAL: NCT00267449
Title: Adjunctive Efficacy Study Of The SoftScan® Optical Breast Imaging System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ART Advanced Research Technologies Inc. (Industry)
Other Study IDs: SSC-311
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-09

CONDITIONS: Breast Cancer
Keywords: Spectroscopy, Near-Infrared; Mammography; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: SoftScan Optical Breast Imaging System

SUMMARY:
The primary study endpoint -SoftScan adjunctive accuracy- will be used to test the hypothesis that the adjunctive combination of the SoftScan with x-ray mammography provides diagnostic accuracy that is significantly better than x-ray mammography alone.

DETAILED DESCRIPTION:
Prospective, serially-recruited, blinded and unblinded, validation study to test that the adjunctive combination of the SoftScan with x-ray mammography provides diagnostic accuracy that is significantly better than x-ray mammography alone. Healthy volunteers and patients scheduled for tissue biopsy/excision of a suspicious breast lesion will be enrolled. Reader Studies will be performed in which interpreting investigators will perform blinded mammography interpretations, and reinterpretations of mammography and SoftScan interpretations. Diagnostic accuracy will be calculated using tissue histopathology as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

Women between the ages of 20 and 80 years of age, who are either healthy or who are scheduled to undergo a tissue biopsy of surgical excision of a suspicious breast lesion for histopathologic diagnosis.

Exclusion Criteria:

For the Healthy Volunteers Population,

* subjects with a history of minor breast procedures involving either breast;
* subjects with a history of major breast procedures involving either breast;
* subjects with a history of significant acute breast abnormalities involving either breast; and
* subjects with a history of significant chronic breast abnormalities involving either breast; and

For Referred For Biopsy Population,

* subjects with a history of minor breast procedures involving either breast that were performed within 6 months prior to enrollment or which have not completed active healing at the time of enrollment;
* subjects with a history of major breast procedures involving either breast;
* subjects with a history of significant acute breast abnormalities involving either breast which have not completed active healing or resolution within 6 months prior to enrollment; and
* subjects with a history of significant chronic breast abnormalities involving either breast.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 950 (Estimated)
Dates: Start 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G Kozikowski, MD, Study Director — ART Advanced Research Technologies Inc.
Locations (6):
- United States (3):
  - University of California-San Diego - Rebecca and John Moores Cancer Center, La Jolla, California
  - Stanford University - Stanford Breast Imaging Center, Stanford, California
  - Martin Memorial Health Systems, Stuart - Robert & Carol Weissman Cancer Center, Stuart, Florida
- Canada (3):
  - CAMIS - Central Alberta Medical Imaging Services, Red Deer, Alberta
  - University Health Network (UNH) - Princess Margaret Hospital, Toronto, Ontario
  - MUHC- McGill University Health Center, Montreal, Quebec

REFERENCES:
- [Background] Intes X. Time-domain optical mammography SoftScan: initial results. Acad Radiol. 2005 Aug;12(8):934-47. doi: 10.1016/j.acra.2005.05.006. PMID 16023382